CLINICAL TRIAL: NCT01780545
Title: The Borealis-2 Clinical Trial: A Randomized Phase 2 Study Comparing Docetaxel Alone to Docetaxel in Combination With OGX-427 in Patients With Relapsed or Refractory Metastatic Urothelial Carcinoma After Receiving a Platinum-containing Regimen: Hoosier Cancer Research Network GU12-160
Brief Title: Phase 2 Study of Docetaxel +/- OGX-427 in Patients With Relapsed or Refractory Metastatic Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Noah Hahn, M.D. (Other)
Collaborators: Achieve Life Sciences (Industry); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor-Investigator, Noah Hahn, M.D., Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GU12-160
Record Dates: First submitted 2013-01-25; First posted 2013-01-31 (Estimated); Results first posted 2017-11-14 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Bladder Cancer; Urothelial Carcinoma
Keywords: OGX-427; Docetaxel
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — apatorsen; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Arm: Arm A (Experimental): Three doses of 600 mg OGX-427 will be administered IV during the loading dose period (days -9 to -1). Following completion of the loading dose period, 600 mg OGX-427 will be given IV weekly on days 1, 8, and 15 of each 21-day cycle.
  Interventions: Drug: OGX-427; Drug: Docetaxel
- Control Arm: Arm B (Active Comparator): Docetaxel (75 mg/M2) will be administered IV on day 1 of each 21 day cycle for a maximum of 10 cycles.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: OGX-427 — Three doses of 600 mg OGX-427 will be administered IV during the loading dose period (days -9 to -1). Following completion of the loading dose period, 600 mg OGX-427 will be given IV weekly on days 1, 8, and 15 of each 21-day cycle. OGX-427 must be administered prior to docetaxel on day 1 of each cycle.
  Following completion of 10 cycles of docetaxel, 600 mg OGX-427 will continue to be administered by IV weekly as maintenance therapy in Arm A participants who do not have disease progression (i.e., stable disease or better). Participants without documented disease progression who have discontinued from study treatment not due to toxicity related to OGX-427 can also continue to receive OGX-427 maintenance as long as they have completed disease assessments following at least 2 cycles of chemotherapy. Maintenance with OGX-427 will continue until disease progression or unacceptable toxicity.
  Arms: Experimental Arm: Arm A
Drug: Docetaxel — For Arm A Only: Docetaxel should be administered immediately following the completion of the OGX-427 infusion.
  For Both Arms: Docetaxel (75 mg/M2) will be administered IV on Day 1 of each 21 day cycle for a maximum of 10 cycles.

SUMMARY:
This is a randomized, open-label Phase 2 clinical trial to evaluate whether suppression of Hsp27 (Heat shock protein 27) production using OGX-427, a second-generation antisense oligonucleotide (ASO), in combination with docetaxel can prolong survival time compared to docetaxel alone in participants with locally advanced or metastatic urothelial carcinoma (UC) that are relapsed or refractory after receiving a platinum-containing regimen.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

Eligible patients will be stratified based on time from prior systemic chemotherapy (< 3 vs ≥ 3 months) and Bellmunt prognostic factors criteria, which include Eastern Cooperative Oncology Group (ECOG) performance status >0, hemoglobin <10g/dL, and presence of liver metastases (0 versus 1-3 risk factors). Within the strata, participants will be randomly assigned with equal probability to either the investigational arm (Arm A: docetaxel + OGX-427) or the control arm (Arm B: docetaxel alone).

INVESTIGATIONAL ARM OGX-427 + DOCETAXEL (Arm A):

LOADING DOSE PERIOD:

Participants randomized onto the investigational arm (Arm A) will receive OGX-427 beginning with a loading dose period prior to the initiation of docetaxel treatment. The first dose of OGX-427 for the loading dose period must be administered within 5 working days of registration and randomization.

During the loading dose period, participants will receive three separate administrations of 600 mg OGX-427 intravenously (IV) (days -9 to -1). There must be at least one "non-infusion" day between each administration of OGX-427 (i.e., every other day) during the loading dose period and between the third loading dose of OGX-427 and day 1 of cycle 1. There should be no more than 7 days between the last loading dose and day 1 of cycle 1.

TREATMENT PERIOD:

During the treatment period, participants randomized to this arm will receive:

* OGX-427 600 mg IV weekly on days 1, 8, and 15 of each 21-day cycle. OGX-427 must be administered prior to docetaxel on day 1 of each cycle.
* Docetaxel (75 mg/M2) IV on day 1 of each 21-day cycle. Docetaxel should be administered immediately following the completion of the OGX-427 infusion.

OGX-427 MAINTENANCE:

Following completion of 10 cycles of docetaxel, 600 mg OGX-427 will continue to be administered by IV weekly as maintenance therapy for participants who do not have disease progression (i.e., stable disease or better). Participants without documented disease progression who have discontinued from study treatment not due to toxicity related to OGX-427 can also continue to receive OGX-427 maintenance as long as they have completed disease assessments following at least 2 cycles of chemotherapy. Maintenance with OGX-427 will continue until disease progression or unacceptable toxicity.

CONTROL ARM - DOCETAXEL ALONE (Arm B):

TREATMENT PERIOD:

During the treatment period, participants randomized to this arm will receive:

- Docetaxel (75 mg/M2) IV on day 1 of each 21-day cycle. The first dose of docetaxel must be administered within 5 working days of registration and randomization. Participants will continue to receive docetaxel on day 1 of each 21-day cycle until disease progression, unacceptable toxicity related to docetaxel, voluntary patient withdrawal, or a maximum of 10 docetaxel cycles.

FOLLOW-UP FOR BOTH ARMS:

Imaging studies will be performed every 6 weeks (i.e., after completion of cycles 2, 4, 6, 8 and 10) until disease progression and with any sign or symptom of new or worsening disease; computed tomography scan (CT) of chest/abdomen/pelvis is preferred but magnetic resonance imaging scan(MRI) is acceptable, especially for participants with increased risk of contrast-related nephropathy or other contraindications. For Arm A, scans will be performed every 2 cycles (6 weeks) +/1 week during the 21-day cycles of docetaxel administration and every 6 weeks during maintenance OGX-427 administration until disease progression; for Arm B, scans will be performed every 6 weeks during the 21-day cycles of docetaxel administration until disease progression. All scans should be completed before the subsequent cycle is scheduled to begin. Bone scans will be repeated, if positive at baseline, every 6 weeks during the first 4 cycles of treatment (i.e., at the end of cycles 2 and 4) and then every 12 weeks thereafter until disease progression (i.e., at the end of cycle 8, at end of treatment, and during maintenance with OGX-427 [Arm A only]).

All participants will have an End of Treatment (EOT) visit when they discontinue study treatment. All participants will be followed until documented disease progression.

Once disease progression is documented, participants will enter a survival follow-up period. All participants must be followed for survival as the primary endpoint. During the survival follow-up period, data will be collected every three months regarding further cancer therapy, secondary malignancy, and survival status.

Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Life Expectancy: Greater than 3 months

Hematopoietic:

* Absolute neutrophil count(ANC)≥ 1,500/mcL
* Hemoglobin ≥ 8 g/dL
* Platelets ≥ 100,000/mcL

Hepatic:

* Bilirubin ≤ 1.1 x upper limit of normal (ULN) (≤ 2.0 x ULN if secondary to Gilbert's disease)
* Aspartate transaminase (AST), serum glutamic oxaloacetic transaminase (SGOT)/alanine transaminase (ALT), serum glutamic pyruvic transaminase (SGPT) ≤ 1.5 X institutional ULN

Renal:

* Serum creatinine ≤ 1.5 x ULN

Cardiac:

* Symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or myocardial infarction within 3 months of randomization.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically documented metastatic or locally inoperable advanced urothelial carcinoma (bladder, urethra, ureter and renal pelvis) (T4b, N2, N3, or M1 disease. NOTE: Aberrant differentiation such as squamous, glandular (adenocarcinoma), and micropapillary are eligible unless the tumor is considered a pure histological variant according to the pathology report. Participants with small cell histology are not eligible.
* Participants must have measurable disease defined as at least one target lesion that has not been irradiated and can be accurately measured in at least one dimension by RECIST v1.1 criteria.
* Participants must have received prior systemic chemotherapy treatment for metastatic urothelial carcinoma. NOTE: Up to 2 prior systemic chemotherapeutic regimens given in the metastatic disease setting for urothelial carcinoma are allowed.
* Specifically, subjects must meet one or more of the following criteria:

  1. Progression during or after treatment with a regimen that includes a platinum salt (e.g., carboplatin or cisplatin) OR
  2. Disease recurrence within one year after neoadjuvant or adjuvant platinum-based systemic chemotherapy, measured from the date of last dose of chemotherapy or surgery until the day the informed consent is signed
* Participants must be ≥18 years since no dosing or adverse event data are currently available on the use of OGX-427 in participants <18 years of age.
* Minimum of 21 days have elapsed since prior major surgery, with recovery from any adverse events.
* Minimum of 14 days have elapsed since any prior radiation therapy, with recovery from any adverse events.
* The effects of OGX-427 on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of treatment with docetaxel in any setting. Participants treated with prior paclitaxel are eligible.
* Prior enrollment in the OncoGenex Phase 2 Study OGX-427-02.
* Participants may not be receiving other investigational agents.
* Participants with known brain or spinal cord metastases are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. NOTE: Brain imaging is not required unless the patient has symptoms or physical signs of central nervous system (CNS) disease.
* History of allergic reactions or severe hypersensitivity reactions to drugs formulated with polysorbate 80 or antisense oligonucleotides.
* Peripheral neuropathy ≥Grade 2.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.
* Cerebrovascular accident or pulmonary embolus within 3 months of randomization.
* Pregnant women and breast feeding women are excluded from this study because of the risk to a fetus due to docetaxel chemotherapy and OGX-427 systemic treatment (fertility toxicology studies have not been completed for OGX-427).
* Active second malignancy (except non-melanomatous skin cancer or incidental prostate cancer found on cystectomy): active secondary malignancy is defined as a current need for cancer therapy or a high possibility (>30%) of recurrence during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-04; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noah Hahn, M.D., Study Chair — Hoosier Cancer Research Network
Locations (35):
- United States (35):
  - University of Alabama Hematology Oncology Clinic at Medical West, Birmingham, Alabama
  - City of Hope: Duarte, Duarte, California
  - City of Hope: Antelope Valley, Lancaster, California
  - USC: Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA: Jonsson Comprehensive Cancer Center, Los Angeles, California
  - IU Health Goshen Hospital, Goshen, Indiana
  - Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Central Indiana Cancer Centers, Indianapolis, Indiana
  - IU Health at Ball Memorial Hospital, Muncie, Indiana
  - University of Maryland: Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University: Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Siteman Cancer Center, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center: Norris Cotton Cancer Center, Manchester, New Hampshire
  - Memorial Sloan-Kettering Cancer Center: Basking Ridge, Basking Ridge, New Jersey
  - John Theurer Cancer Center: Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of New Mexico Cancer Center: Albuquerque, Albuquerque, New Mexico
  - University of New Mexico Cancer Center: Las Cruces, Las Cruces, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan-Kettering Cancer Center: Commack, Commack, New York
  - New York University Clinical Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center: Main Campus, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Memorial Sloan-Kettering Cancer Center: Rockville Centre, Rockville Centre, New York
  - Memorial Sloan-Kettering Cancer Center: Sleepy Hollow, Sleepy Hollow, New York
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Cleveland Clinic: Taussig Cancer Institute, Cleveland, Ohio
  - Lake Health: University Hospitals Seidman Cancer Center, Mentor, Ohio
  - UHHS Chagrin Highlands: Seidman Cancer Center, Orange, Ohio
  - Thomas Jefferson University: Kimmel Cancer Center, Philadelphia, Pennsylvania
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Jonathan E. Rosenberg, Noah M. Hahn, Meredith M. Regan, Cindy Jacobs, Patricia S. Stewart, Toni K. Choueiri. The Borealis-2 clinical trial: A randomized phase II study of OGX-427 plus docetaxel versus docetaxel alone in relapsed/refractory metastatic urothelial cancer. J Clin Oncol 31, 2013 (suppl; abstr TPS4588^) http://abstracts2.asco.org/AbstView_132_114639.html
- [Background] Choueiri TK, Hahn NM, Pal SK, Alva AS, Dreicer R, Starodub A, Sonpavde G, Hoffman-Censits JH, Picus J, Balar AV, Guancial EA, Regan MM, Jacobs C, Stewart PS, Rosenberg JE. The Borealis-2 clinical trial: A randomized phase 2 study of OGX-427 (apatorsen) plus docetaxel versus docetaxel alone in relapsed/refractory metastatic urothelial cancer. J Clin Oncol 32:5s, 2014 (suppl; abstr TPS4593^)
- [Background] Choueiri TK, Hahn NM, Alva AS, Lauer RC, Dreicer R, Picus J, Pili R, Balar AV, Sonpavde G, Hoffman-Censits JH, Guancial EA, Alter R, Regan MM, Jacobs C, Stewart PS, Pal SK, Rosenberg JE. The Borealis-2 clinical trial: A randomized phase 2 study of OGX-427 (Apatorsen) plus docetaxel versus docetaxel alone in relapsed/refractory metastatic urothelial cancer. J Clin Oncol 33:5s, 2015 (suppl; abstr TPS4577)
- See also: Hoosier Cancer Research Network Website — http://www.hoosiercancer.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Arm: Arm A: Three doses of 600 mg OGX-427 will be administered IV during the loading dose period (days -9 to -1). Following completion of the loading dose period, 600 mg OGX-427 will be given IV weekly on days 1, 8, and 15 of each 21-day cycle. OGX-427 must be administered prior to docetaxel on day 1 of each cycle.
  Following completion of 10 cycles of docetaxel, 600 mg OGX-427 will continue to be administered by IV weekly as maintenance therapy in Arm A participants who do not have disease progression (i.e., stable disease or better). Maintenance with OGX-427 will continue until disease progression or unacceptable toxicity.
  Docetaxel: For Arm A Only: Docetaxel should be administered immediately following the completion of the OGX-427 infusion.
  For Both Arms: Docetaxel (75 mg/M2) will be administered IV on Day 1 of each 21 day cycle for a maximum of 10 cycles.
- Control Arm: Arm B: Docetaxel (75 mg/M2) will be administered IV on day 1 of each 21 day cycle for a maximum of 10 cycles.
  Docetaxel: For Arm A Only: Docetaxel should be administered immediately following the completion of the OGX-427 infusion.
  For Both Arms: Docetaxel (75 mg/M2) will be administered IV on Day 1 of each 21 day cycle for a maximum of 10 cycles.
Period: Overall Study
Arm/Group | Experimental Arm: Arm A | Control Arm: Arm B
Started | 99 | 101
Completed | 95 | 99
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Arm: Arm A | Control Arm: Arm B | Total
Number analyzed (Participants) | 99 | 101 | 200
Age, Continuous [Median (Full Range); unit: years] | 68 [43 to 90] | 67 [35 to 92] | 67 [35 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 74 | 75 | 149
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 94 | 98 | 192
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 89 | 92 | 181
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: To determine whether docetaxel administered in combination with OGX-427 provides a survival benefit compared to docetaxel alone.
Time Frame: 36 Months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental Arm: Arm A | Control Arm: Arm B
Number analyzed (Participants) | 99 | 101
months | 6.4 [4.6 to 9.2] | 5.9 [4.8 to 7.3]

2. Secondary Outcome: Safety and Toxicity of Regimen
Description: To compare the safety and toxicity of OGX-427 in combination with docetaxel to that of docetaxel alone. A summary of per-patient maxiumy grade adverse events of any type is included in the Outcome Measure. Full adverse event information will be submitted further in the record.
Time Frame: 36 Months
Population: 190 participants who intiated protocol treatment were included in the safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Arm: Arm A | Control Arm: Arm B
Number analyzed (Participants) | 94 | 96
Participants
  Maximum AE Grade: 0 | 0 | 2
  Maximum AE Grade: 1 | 6 | 7
  Maximum AE Grade: 2 | 11 | 15
  Maximum AE Grade: 3 | 40 | 41
  Maximum AE Grade: 4 | 32 | 26
  Maximum AE Grade: 5 | 5 | 6

3. Secondary Outcome: Overall Response Rate
Description: To compare overall response rate (ORR) between the treatment arms.
Time Frame: Every 6 weeks
Population: Data for this secondary outcome measure was not collected nor analyzed.
Arm/Group | Experimental Arm: Arm A | Control Arm: Arm B
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Survival (OS) According to Baseline Serum Hsp27 Level.
Description: A subgroup analysis to determine the median overall survival time based on baseline Hsp27 levels.
Time Frame: 36 months
Population: Subjects with a baseline Hsp27 level were included in this subgroup analysis
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Hsp27 <5.7ng/mL: Subjects with a baseline Hsp27 level <5.7 ng/mL
- Hsp27 >=5.7ng/mL: Subjects with a baseline Hsp27 level >=5.7 ng/mL
Arm/Group | Hsp27 <5.7ng/mL | Hsp27 >=5.7ng/mL
Number analyzed (Participants) | 79 | 82
months | 9.4 [5.8 to 12.4] | 4.7 [3.7 to 6.0]

5. Secondary Outcome: Hsp27 Expression in Archival Tissue
Description: To evaluate the association of urothelial carcinoma expression of Hsp27 measured by immunohistochemistry (IHC) in archival tissue with clinical outcomes.
Time Frame: Cycle 1
Population: Data for this secondary outcome was not collected or analyzed.
Groups:
- Experimental Arm: Arm A: Three doses of 600 mg OGX-427 will be administered IV during the loading dose period (days -9 to -1). Following completion of the loading dose period, 600 mg OGX-427 will be given IV weekly on days 1, 8, and 15 of each 21-day cycle.
  OGX-427: Three doses of 600 mg OGX-427 will be administered IV during the loading dose period (days -9 to -1). Following completion of the loading dose period, 600 mg OGX-427 will be given IV weekly on days 1, 8, and 15 of each 21-day cycle. OGX-427 must be administered prior to docetaxel on day 1 of each cycle.
  Following completion of 10 cycles of docetaxel, 600 mg OGX-427 will continue to be administered by IV weekly as maintenance therapy in Arm A participants who do not have disease progression (i.e., stable disease or better). Participants without documented disease progression who have discontinued from study treatment not due to toxicity related to OGX-427 can also continue to receive OGX-427 maintenance as long as they have completed disease
Arm/Group | Experimental Arm: Arm A | Control Arm: Arm B
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Effect of Therapy Regimen on Circulating Tumor Cells (CTCs)and Correlative Analysis of Telomerase Activity
Description: To evaluate the effect of therapy with docetaxel and OGX-427 on peripheral blood circulating tumor cells (CTCs) enumeration and expression of Hsp27 and other relevant proteins via immunoflourescence, and levels of telomerase by quantitative polymerase chain reaction (PCR), and explore their relation with clinical outcomes.
Time Frame: Prior to screening, prior to first loading dose, and prior to cycles 1, 2, 3 and 5
Population: Data for this secondary objective was not collected or analyzed.
Arm/Group | Experimental Arm: Arm A | Control Arm: Arm B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Duration of study, up to 36 months
Arm/Group | Experimental Arm: Arm A | Control Arm: Arm B
All-Cause Mortality (participants affected / at risk) | 78/99 | 86/101
Serious Adverse Events (participants affected / at risk) | 56/99 | 45/101
Other Adverse Events (participants affected / at risk) | 94/99 | 93/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm: Arm A (N=99) | Control Arm: Arm B (N=101)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 4 (5) | 3 (3)
APPENDICITIS (Infections and infestations) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ASCITES (Gastrointestinal disorders) | 1 (2) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 1 (1)
BLADDER PERFORATION (Renal and urinary disorders) | 1 (1) | 0 (0)
CATHETER RELATED INFECTION (Infections and infestations) | 2 (2) | 0 (0)
CHILLS (General disorders) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 2 (2) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 1 (2)
CREATININE INCREASED (Investigations) | 1 (1) | 0 (0)
DEATH NOS (General disorders) | 1 (1) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 6 (6) | 4 (5)
DELIRIUM (Psychiatric disorders) | 1 (1) | 0 (0)
DUODENAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 6 (7) | 8 (8)
FEVER (General disorders) | 7 (8) | 1 (1)
GASTRIC HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 1 (1) | 1 (1)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS (General disorders) | 1 (1) | 0 (0)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 1 (1) | 1 (1)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 4 (4) | 3 (4)
INTRACRANIAL HEMORRHAGE (Nervous system disorders) | 1 (1) | 1 (1)
LUNG INFECTION (Infections and infestations) | 2 (3) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 1 (1) | 0 (0)
MULTI-ORGAN FAILURE (General disorders) | 1 (1) | 0 (0)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 2 (2) | 0 (0)
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
RENAL AND URINARY DISORDERS (Renal and urinary disorders) | 2 (2) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
SEIZURE (Nervous system disorders) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 13 (13) | 7 (7)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 (3) | 2 (2)
STROKE (Nervous system disorders) | 1 (1) | 0 (0)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1) | 2 (2)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 10 (13) | 4 (4)
VASCULAR DISORDERS (Vascular disorders) | 1 (1) | 1 (1)
VOMITING (Gastrointestinal disorders) | 2 (2) | 2 (2)
ABDOMINAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 1 (1)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 1 (1)
CATARACT (Eye disorders) | 0 (0) | 1 (2)
COLONIC FISTULA (Gastrointestinal disorders) | 0 (0) | 1 (1)
COLONIC PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 0 (0) | 2 (2)
EDEMA LIMBS (General disorders) | 0 (0) | 1 (1)
FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HEMATOMA (Vascular disorders) | 0 (0) | 1 (1)
HEPATIC FAILURE (Hepatobiliary disorders) | 0 (0) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (2)
KIDNEY INFECTION (Infections and infestations) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
PAIN (General disorders) | 0 (0) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 1 (1)
PERICARDIAL TAMPONADE (Cardiac disorders) | 0 (0) | 1 (1)
PERIPHERAL ISCHEMIA (Vascular disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
SINUSITIS (Infections and infestations) | 0 (0) | 1 (1)
SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1)
SMALL INTESTINE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
WOUND INFECTION (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm: Arm A (N=99) | Control Arm: Arm B (N=101)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 (2) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 28 (40) | 13 (15)
ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 3 (4) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 1 (1)
AKATHISIA (Nervous system disorders) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 10 (14) | 7 (8)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 6 (8) | 6 (7)
ALLERGIC REACTION (Immune system disorders) | 2 (2) | 3 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 26 (30) | 26 (28)
ANEMIA (Blood and lymphatic system disorders) | 38 (88) | 36 (77)
ANOREXIA (Metabolism and nutrition disorders) | 42 (69) | 30 (36)
ANXIETY (Psychiatric disorders) | 4 (4) | 7 (7)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 9 (11) | 4 (6)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 6 (9) | 8 (10)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 (2) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 11 (14) | 20 (24)
BLADDER SPASM (Renal and urinary disorders) | 1 (1) | 0 (0)
BLOATING (Gastrointestinal disorders) | 4 (4) | 1 (2)
BLOOD AND LYMPHATIC SYSTEM DISORDERS (Blood and lymphatic system disorders) | 3 (3) | 3 (4)
BLOOD BILIRUBIN INCREASED (Investigations) | 3 (3) | 1 (1)
BLURRED VISION (Eye disorders) | 4 (4) | 5 (6)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (9)
BRONCHIAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
BRONCHOPULMONARY HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
BRUISING (Injury, poisoning and procedural complications) | 3 (4) | 2 (2)
BULLOUS DERMATITIS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
BUTTOCK PAIN (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
CARDIAC DISORDERS (Cardiac disorders) | 1 (1) | 5 (5)
CATHETER RELATED INFECTION (Infections and infestations) | 1 (1) | 0 (0)
CD4 LYMPHOCYTES DECREASED (Investigations) | 1 (3) | 1 (1)
CHEST PAIN - CARDIAC (Cardiac disorders) | 1 (1) | 2 (2)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
CHILLS (General disorders) | 24 (27) | 12 (13)
CHOLESTEROL HIGH (Investigations) | 2 (2) | 5 (5)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 3 (6) | 0 (0)
CONFUSION (Psychiatric disorders) | 4 (4) | 4 (5)
CONJUNCTIVITIS (Eye disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 37 (49) | 25 (29)
COUGH (Respiratory, thoracic and mediastinal disorders) | 18 (32) | 15 (17)
CREATININE INCREASED (Investigations) | 30 (46) | 12 (19)
CUSHINGOID (Endocrine disorders) | 1 (2) | 0 (0)
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 1 (1) | 3 (3)
CYTOKINE RELEASE SYNDROME (Immune system disorders) | 2 (2) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 15 (15) | 10 (10)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 2 (2) | 0 (0)
DEPRESSION (Psychiatric disorders) | 4 (4) | 5 (5)
DIARRHEA (Gastrointestinal disorders) | 47 (72) | 35 (60)
DIZZINESS (Nervous system disorders) | 14 (14) | 11 (11)
DRY EYE (Eye disorders) | 3 (3) | 1 (1)
DRY MOUTH (Gastrointestinal disorders) | 2 (2) | 3 (3)
DRY SKIN (Skin and subcutaneous tissue disorders) | 11 (11) | 10 (10)
DYSGEUSIA (Nervous system disorders) | 17 (22) | 17 (20)
DYSPEPSIA (Gastrointestinal disorders) | 5 (5) | 5 (5)
DYSPHAGIA (Gastrointestinal disorders) | 4 (4) | 3 (3)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 28 (35) | 29 (35)
EAR AND LABYRINTH DISORDERS (Ear and labyrinth disorders) | 1 (1) | 1 (1)
EDEMA FACE (General disorders) | 2 (3) | 2 (3)
EDEMA LIMBS (General disorders) | 21 (33) | 25 (41)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 4 (6)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
ERYTHRODERMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
EYE DISORDERS (Eye disorders) | 4 (7) | 5 (8)
EYE PAIN (Eye disorders) | 1 (1) | 1 (1)
FACIAL PAIN (General disorders) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 5 (5) | 5 (8)
FATIGUE (General disorders) | 63 (119) | 66 (128)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
FEVER (General disorders) | 28 (36) | 14 (19)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 9 (10) | 3 (3)
FLATULENCE (Gastrointestinal disorders) | 2 (2) | 2 (2)
FLU LIKE SYMPTOMS (General disorders) | 6 (6) | 1 (1)
FLUSHING (Vascular disorders) | 3 (3) | 3 (3)
GAIT DISTURBANCE (General disorders) | 2 (2) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 5 (5) | 1 (1)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 12 (17) | 3 (7)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS (General disorders) | 5 (17) | 4 (5)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 17 (22) | 17 (21)
GENITAL EDEMA (Reproductive system and breast disorders) | 4 (6) | 1 (3)
GLAUCOMA (Eye disorders) | 1 (1) | 0 (0)
GLUCOSE INTOLERANCE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HALLUCINATIONS (Psychiatric disorders) | 2 (2) | 2 (2)
HEADACHE (Nervous system disorders) | 11 (16) | 7 (12)
HEARING IMPAIRED (Ear and labyrinth disorders) | 3 (3) | 2 (2)
HEMATOMA (Vascular disorders) | 1 (1) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 9 (11) | 10 (12)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (7)
HOT FLASHES (Vascular disorders) | 4 (4) | 0 (0)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 4 (7) | 7 (11)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 18 (45) | 14 (22)
HYPERKALEMIA (Metabolism and nutrition disorders) | 7 (16) | 6 (8)
HYPERMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
HYPERNATREMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 12 (18) | 13 (15)
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
HYPERURICEMIA (Metabolism and nutrition disorders) | 3 (9) | 4 (4)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 14 (27) | 15 (21)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 8 (11) | 7 (12)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 9 (15) | 3 (3)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 23 (32) | 11 (16)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 12 (18) | 12 (19)
HYPOTENSION (Vascular disorders) | 8 (11) | 7 (8)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 7 (13) | 3 (5)
INFUSION RELATED REACTION (General disorders) | 7 (9) | 1 (1)
INR INCREASED (Investigations) | 7 (13) | 3 (3)
INSOMNIA (Psychiatric disorders) | 11 (12) | 19 (24)
INTRAOPERATIVE MUSCULOSKELETAL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 1 (3) | 0 (0)
LETHARGY (Nervous system disorders) | 1 (2) | 0 (0)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 2 (3) | 4 (4)
LOCALIZED EDEMA (General disorders) | 2 (2) | 3 (4)
LYMPHOCYTE COUNT DECREASED (Investigations) | 17 (58) | 11 (34)
LYMPHOCYTE COUNT INCREASED (Investigations) | 1 (2) | 0 (0)
MALAISE (General disorders) | 4 (4) | 1 (1)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1) | 3 (3)
METABOLISM AND NUTRITION DISORDERS (Metabolism and nutrition disorders) | 3 (5) | 3 (4)
MUCOSAL INFECTION (Infections and infestations) | 2 (2) | 3 (3)
MUCOSITIS ORAL (Gastrointestinal disorders) | 15 (26) | 21 (26)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (4)
MUSCLE WEAKNESS RIGHT-SIDED (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER (Musculoskeletal and connective tissue disorders) | 11 (16) | 6 (6)
MYALGIA (Musculoskeletal and connective tissue disorders) | 6 (8) | 6 (12)
NAIL DISCOLORATION (Skin and subcutaneous tissue disorders) | 7 (10) | 7 (7)
NAIL RIDGING (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 3 (5)
NAUSEA (Gastrointestinal disorders) | 41 (63) | 34 (49)
NECK EDEMA (General disorders) | 1 (1) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
NERVOUS SYSTEM DISORDERS (Nervous system disorders) | 2 (2) | 2 (2)
NEUTROPHIL COUNT DECREASED (Investigations) | 35 (58) | 33 (46)
NON-CARDIAC CHEST PAIN (General disorders) | 7 (7) | 2 (2)
ORAL DYSESTHESIA (Gastrointestinal disorders) | 1 (1) | 1 (1)
ORAL PAIN (Gastrointestinal disorders) | 3 (3) | 2 (5)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTITIS EXTERNA (Infections and infestations) | 1 (1) | 0 (0)
PAIN (General disorders) | 19 (27) | 20 (27)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 14 (27) | 16 (23)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
PAPULOPUSTULAR RASH (Infections and infestations) | 1 (1) | 0 (0)
PARESTHESIA (Nervous system disorders) | 2 (2) | 2 (7)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (3) | 6 (8)
PENILE PAIN (Reproductive system and breast disorders) | 2 (3) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1) | 0 (0)
PERINEAL PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 3 (4) | 7 (9)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 28 (46) | 22 (28)
PHLEBITIS (Vascular disorders) | 1 (1) | 0 (0)
PHOTOPHOBIA (Eye disorders) | 1 (1) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 12 (16) | 10 (13)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 1 (1) | 1 (1)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
POSTOPERATIVE HEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
PROTEINURIA (Renal and urinary disorders) | 4 (4) | 1 (3)
PRURITUS (Skin and subcutaneous tissue disorders) | 11 (19) | 8 (10)
PSYCHIATRIC DISORDERS (Psychiatric disorders) | 1 (1) | 1 (1)
PURPURA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 13 (22) | 8 (9)
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 1 (3)
RENAL AND URINARY DISORDERS (Renal and urinary disorders) | 7 (11) | 7 (14)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (6)
RESTLESSNESS (Psychiatric disorders) | 2 (2) | 0 (0)
RHINITIS INFECTIVE (Infections and infestations) | 2 (2) | 3 (3)
SCALP PAIN (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
SINUS BRADYCARDIA (Cardiac disorders) | 1 (1) | 1 (1)
SINUS DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 8 (9) | 5 (6)
SINUSITIS (Infections and infestations) | 1 (1) | 2 (2)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS (Skin and subcutaneous tissue disorders) | 13 (25) | 7 (12)
SKIN INFECTION (Infections and infestations) | 3 (3) | 3 (4)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 5 (5)
STOMACH PAIN (Gastrointestinal disorders) | 1 (1) | 2 (2)
SURGICAL AND MEDICAL PROCEDURES (Surgical and medical procedures) | 2 (2) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 3 (4)
TESTICULAR PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0)
THROMBOEMBOLIC EVENT (Vascular disorders) | 7 (7) | 5 (7)
TINNITUS (Ear and labyrinth disorders) | 4 (4) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 0 (0)
TUMOR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 0 (0)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 2 (3) | 1 (2)
URINARY FREQUENCY (Renal and urinary disorders) | 8 (9) | 12 (13)
URINARY INCONTINENCE (Renal and urinary disorders) | 5 (8) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 15 (28) | 11 (12)
URINARY TRACT PAIN (Renal and urinary disorders) | 2 (2) | 1 (1)
URINARY URGENCY (Renal and urinary disorders) | 1 (1) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
VOICE ALTERATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
VOMITING (Gastrointestinal disorders) | 20 (23) | 16 (27)
WATERING EYES (Eye disorders) | 4 (6) | 5 (6)
WEIGHT GAIN (Investigations) | 2 (4) | 0 (0)
WEIGHT LOSS (Investigations) | 13 (17) | 15 (18)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
WHITE BLOOD CELL DECREASED (Investigations) | 31 (54) | 23 (35)
WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0)
AGITATION (Psychiatric disorders) | 0 (0) | 1 (1)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
APNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BLADDER INFECTION (Infections and infestations) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (2)
CONCENTRATION IMPAIRMENT (Nervous system disorders) | 0 (0) | 1 (1)
DELIRIUM (Psychiatric disorders) | 0 (0) | 1 (1)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 2 (2)
EDEMA TRUNK (General disorders) | 0 (0) | 3 (3)
ENDOCRINE DISORDERS - OTHER, SPECIFY (Endocrine disorders) | 0 (0) | 1 (1)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 (0) | 1 (1)
FECAL INCONTINENCE (Gastrointestinal disorders) | 0 (0) | 1 (1)
FLASHING LIGHTS (Eye disorders) | 0 (0) | 1 (1)
HEMOGLOBIN INCREASED (Investigations) | 0 (0) | 1 (2)
HEMOLYTIC UREMIC SYNDROME (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
HEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 2 (2)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
INJECTION SITE REACTION (General disorders) | 0 (0) | 1 (1)
LARYNGEAL HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
LARYNGEAL MUCOSITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
LIP INFECTION (Infections and infestations) | 0 (0) | 2 (2)
LIP PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
LOWER GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
LUNG INFECTION (Infections and infestations) | 0 (0) | 2 (2)
LYMPHEDEMA (Vascular disorders) | 0 (0) | 2 (2)
NAIL LOSS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ORAL HEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
PAPILLEDEMA (Eye disorders) | 0 (0) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
RECTAL FISTULA (Gastrointestinal disorders) | 0 (0) | 1 (1)
RECTAL PAIN (Gastrointestinal disorders) | 0 (0) | 3 (4)
SCROTAL PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 1 (1)
TREMOR (Nervous system disorders) | 0 (0) | 2 (2)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 2 (2)
URINE DISCOLORATION (Renal and urinary disorders) | 0 (0) | 1 (1)
URINE OUTPUT DECREASED (Investigations) | 0 (0) | 1 (1)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VAGINAL HEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (6)
VASCULAR DISORDERS - OTHER, SPECIFY (Vascular disorders) | 0 (0) | 1 (1)
VITREOUS HEMORRHAGE (Eye disorders) | 0 (0) | 1 (2)
WOLFF-PARKINSON-WHITE SYNDROME (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT01780545/Prot_SAP_000.pdf